CLINICAL TRIAL: NCT07242274
Title: A Multicenter, Randomized, Open-Label, Phase 3 Study Evaluating the Efficacy and Safety of JMKX001899 Versus Docetaxel in Previously Treated Patients With KRAS G12C-Mutant Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Phase 3 Trial of JMKX001899 Versus Docetaxel in Previously Treated Advanced or Metastatic KRAS G12C-Mutant NSCLC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jemincare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JY-JM1899-103
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: NSCLC (Non-small Cell Lung Cancer)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JMKX001899 (Experimental): Orally, once daily
  Interventions: Drug: JMKX001899
- Docetaxel (Active Comparator): By IV infusion every 21 days
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: JMKX001899 — Orally, once daily
  Arms: JMKX001899
Drug: Docetaxel — By IV infusion every 21 days
  Arms: Docetaxel

SUMMARY:
This is a multicenter, randomized, open-label, phase 3 clinical trial designed to evaluate the efficacy and safety of JMKX001899 compared to docetaxel in patients with previously treated, KRAS G12C-mutant advanced or metastatic non-small cell lung cancer (NSCLC).

KRAS G12C mutation is present in a subset of NSCLC patients. While docetaxel is a standard chemotherapy option, JMKX001899 is an investigational, targeted therapy designed to selectively inhibit the KRAS G12C mutation. This trial aims to determine whether JMKX001899 offers a superior clinical benefit compared to standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Histologically or cytologically confirmed NSCLC.
3. Failure of at least one prior line of therapy for locally advanced/metastatic disease, that included a platinum-based chemotherapy and a PD-1/PD-L1 inhibitor.
4. At least one measurable lesion as defined by RECIST version 1.1.

Exclusion Criteria:

1. Known concomitant presence of other oncogenic driver mutations or rearrangements with established targeted therapies .
2. Previous treatment with any KRAS G12C-targeted agent.
3. Prior docetaxel therapy in the locally advanced/metastatic setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 1 year
  Progression-Free Survival

SECONDARY OUTCOMES:
OS | 3 years
  Overall Survival
AE | from first dose to 28 days after the last dose
  Adverse Event

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, Doctor, Principal Investigator — Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No